CLINICAL TRIAL: NCT04761926
Title: Investigating Hearing With the Ponto 4, a Bone Anchored Hearing Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BC110
Record Dates: First submitted 2021-01-20; First posted 2021-02-21 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hearing Loss, Conductive; Hearing Loss, Mixed
Keywords: Hearing loss; hearing disorder,; ear diseases; BAHS
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Hearing Loss; Hearing Disorders; Ear Diseases | interventions — Audiometry; Patient Reported Outcome Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm (Experimental): Asessments for the hearing with Ponto 4 sound processor on the implanted ear(s).
  Interventions: Device: Audiometry

INTERVENTIONS:
Device: Audiometry — Audiometry: Thresholds from the audiogram obtained when Ponto 4 were fitted. Pure tone air conduction (AC) and bone conduction (BC) audiometry conducted at the visit.
  Speech recognition in quiet: Speech intelligibility is measured in a soundproof room using the Matrix sentences presented from a loudspeaker. The Matrix test includes five-word sentences with a fixed syntactical structure and limited contextual cues. A list of 20 sentences is compiled from these words, ensuring that no sentence is repeated twice. This test will be obtained both unaided and aided (with and without the Ponto 4(s)).
  Sound field Audiometry: Detection of sound field thresholds presented from a loudspeaker. Thresholds will be obtained both unaided and aided and the test order will be balanced between subjects. During these measurements, the Ponto 4 will be programmed in omni-directional mode, with noise reduction and feedback management system turned off.
  Other Names: Speach recognition in quiet; Sound field audiometry; Patient reported outcomes

SUMMARY:
The study is a combined retrospective (fitting visit) and prospective (study visit), multi-center, single arm study The study is part of the Post Market Clinical Follow (PMCF) activity. The investigational device used in this study is the Ponto 4 already fitted to the subjects prior to the study. The device is CE marked and available on the market since June 2019.

Treatment is not provided in the study therefore risks are limited to the audiological measurements. The audiological measurements in the study are standard non-invasive measurements already familiar to the clinics.

The hearing with Ponto 4 will be evaluated via speech and hearing tests, and patient reported outcomes.

DETAILED DESCRIPTION:
This is a post market clinical follow up (PMCF) study with the purpose of gather knowledge on the use and performance of the Ponto 4 device on existing Ponto 4 users. The study does not include any treatment or fitting of new devices, instead the real-life application of the use of Ponto 4 on subjects already using Ponto 4(s) are investigated.

The Investigational Device used in the study is Ponto 4, a CE marked, and FDA cleared bone anchored hearing solution, produced by Oticon Medical AB and commercially available since June 2019.

The recruitment for this clinical investigation will be performed among subjects who have already received a Ponto 4 device as a minimum 1.5 month prior to the study. 20 patients, including minors down to 12 years old, with a conductive, mixed hearing loss or single-sided deafness will be included. The rationale for including minors is that they are also users of the device, and it is found important to collect data from their experience of using the device as well.

The study is a retrospective and prospective, multi-center study. It has one visit of 2,5-3 hours for adult subjects ≥18 years old. To minimize the burden and risks of tiredness for the minor subjects from 12-17 years old, the protocol activities can be divided into two visits. The decision will be based on the Investigators discretion.

The majority of the objectives of the study are prospectively collected whereas the BC In-situ (hearing with the Ponto 4 on) and audiometric data from the time of the fitting of Ponto 4, are collected retrospectively from the time of the fitting of Ponto 4 (aka the fitting visit).

The overall objectives of the study are to investigate the improvement in hearing with the Ponto 4(s) on the implanted ear(s), in terms of the subject's ability to hear sounds and understand speech when using the device.

The primary endpoint is to investigate the improvement in hearing with the Ponto 4(s) on the implanted ear for patients within intended use.

These will be evaluated through a hearing and a speech test, both assessing the hearing with the Ponto 4(s) both on and off. Additionally, the subject will complete 2 patient reported outcome, report daily usage time of the device and assess satisfaction of connectivity devices.

Minimal risks are expected for subjects participating in the study. Treatment is not provided in the study therefore risks are limited to the audiological measurements. The audiological measurements in the study are standard non-invasive measurements already familiar to the clinics. The measurements will require an extra effort and may be found slightly tiring by the subject. To mitigate the risk of tiredness the subject will be given the opportunity to have breaks during the visit.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. 12 years old and above
3. Subjects with hearing loss fitted unilaterally or bilaterally with the Ponto 4(s) on abutment at least 1.5 months prior to being enrolled in the study
4. Fluent in local language, as judged by the investigator

Exclusion Criteria:

1. Participation in another clinical investigation which might cause interference with study participation.
2. Subjects who do not have the ability or are un-willing to follow investigational procedures/requirements, e.g. to complete patient related outcome (PRO's) according to investigators discretion

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris L Jacobsen, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ponto 4 Sound Processor Users: Asessments for the hearing with Ponto 4 sound processor on the implanted ear(s).
  Audiometry: Audiometry: Thresholds from the audiogram obtained when Ponto 4 were fitted. Pure tone air conduction (AC) and bone conduction (BC) audiometry conducted at the visit.
  Speech recognition in quiet: Speech intelligibility is measured in a soundproof room using the Matrix sentences presented from a loudspeaker. The Matrix test includes five-word sentences with a fixed syntactical structure and limited contextual cues. A list of 20 sentences is compiled from these words, ensuring that no sentence is repeated twice. This test will be obtained both unaided and aided (with and without the Ponto 4(s)).
  Sound field Audiometry: Detection of sound field thresholds presented from a loudspeaker. Thresholds will be obtained both unaided and aided and the test order will be balanced between subjects. During these measurements, the Ponto 4 will be programmed in omni-directional mode, with noise reduction and feedback management system turned off.
Period: Overall Study
Arm/Group | Ponto 4 Sound Processor Users
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ponto 4 Sound Processor Users
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (17.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: To Investigate the Improvement in Hearing With the Ponto 4 (s) on the Implanted Ear for Patients Within Intended Use.
Description: Functional gain with Ponto 4, i.e. the difference between average unaided and aided sound field thresholds. The functional gain (PTA4) is calculated as the average of frequencies 500, 1000, 2000 and 4000 Hz.
Time Frame: The outcome measure was assessed during Study Visit 1 (Day 1).
Population: only 18 subjects had measurable thresholds for all 4 frequencies to be calculated for the PTA4 of functional gain.
Measure: Mean (Standard Deviation); unit: [dB]
Arm/Group | Ponto 4 Sound Processor Users
Number analyzed (Participants) | 18
[dB] | 31.5 (9.5)

2. Secondary Outcome: B. To Assess the Improvement of Hearing With the Ponto 4 on the Implanted Ear(s).
Description: 1. Functional gain with Ponto 4, i.e. the difference between unaided and aided sound field thresholds, for frequencies 250, 500, 1000, 2000, 3000, 4000, 6000 and 8000 Hz.
Time Frame: The outcome measure was assessed during Study Visit 1 (Day 1).
Measure: Mean (Standard Deviation); unit: [dB]
Arm/Group | Ponto 4 Sound Processor Users
Number analyzed (Participants) | 19
[dB]
  250Hz | 14.2 (9.9)
  500Hz | 28.7 (12.0)
  1000Hz | 36.6 (9.9)
  2000Hz | 28.6 (13.8)
  3000Hz | 32.9 (11.6)
  4000Hz | 32.8 (8.6)
  6000Hz | 22.7 (10.2)
  8000Hz | 22.1 (12.3)

3. Secondary Outcome: C. To Assess the Improvement of Speech Recognition With Ponto 4 on the Implanted Ear(s).
Description: Difference in speech recognition score in percent between unaided and aided, assessed in quiet.
  Speech recognition was measured in free field using the Matrix sentences test. The Matrix test includes five-word sentences with a fixed syntactical structure and limited contextual cues. A formula selects a word from a category (name, verb, number, adjective and noun) and creates a five-word sentence. A word from each category is chosen at random to create the sentence. A list of 20 sentences is compiled from these words, ensuring that no sentence is repeated twice.
  Speech was presented from a loudspeaker 1 meter in front of the subject (0 degree azimuth). The speech signal was fixed at 65 dB SPL (C-weighted). The subject had to repeat as many words as possible after each sentence. For the aided condition, Ponto 4 was tested in the subject's user settings. The test order of aided and unaided condition was balanced across subjects.
Time Frame: The outcome measure was assessed during Study Visit 1 (Day 1).
Measure: Mean (Standard Deviation); unit: percentage points (% points)
Arm/Group | Ponto 4 Sound Processor Users
Number analyzed (Participants) | 19
percentage points (% points) | 55.9 (31.7)

4. Secondary Outcome: G. To Assess the Degree to Which the Ponto 4 Compensates for the BC Hearing Loss on the Implanted Ear(s).
Description: 1. Effective gain defined as the difference in dB between aided sound field thresholds with Ponto 4, and BC In-situ thresholds on the aided ear(s) measured at the time of the fitting of Ponto 4(s). The effective gain is calculated for frequencies 250, 500, 1000, 2000, 3000, 4000, 6000 and 8000 Hz.
Time Frame: The assessment for this outcome measure was based on the BC in situ test conducted during a visit at least 6 weeks prior to Study Visit 1 (data collected retrospectively), and an aided sound field thresholds test conducted on Study Visit Day 1.
Population: Ponto 4 Sound Processor Users
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Ponto 4 Sound Processor Users
Number analyzed (Participants) | 14
dB
  250Hz | 22.0 (7.3)
  500Hz | 7.14 (7.84)
  1000Hz | 3.21 (7.69)
  2000Hz | 2.86 (8.25)
  3000Hz | 10.20 (7.0)
  4000Hz | 13.8 (7.1)
  6000Hz | 17.0 (9.4)
  8000Hz | 12.3 (9.7)

5. Secondary Outcome: H. To Evaluate the Above Objectives on Individual Levels
Description: Endpoints A1, B1, C1 analyzed as the proportion of subjects whose performance improved or remained the same (difference ≥ 0) in unaided to aided comparisons.
Time Frame: The outcome measure was assessed during Study Visit 1 (Day 1).
Measure: Number; unit: Percentage of participants (%)
Arm/Group | Ponto 4 Sound Processor Users
Number analyzed (Participants) | 19
Percentage of participants (%)
  PTA4 unaided to aided condition | 100
  All individual frequencies unaided to aided condition | 100
  Speech recognition scores unaided to aided condition | 100

6. Secondary Outcome: I. To Assess the Degree of Inner Ear Hearing Loss Degradation on the Implanted Ear(s) (for SSD the Stimulated Ear).
Description: 1. Hearing loss degradation is the difference in dB between masked (if not available unmasked) BC thresholds obtained at the study visit, and at the visit when Ponto 4(s) was fitted.
  Hearing loss degradation for subjects with MHL/CHL is the difference in dB between masked (if not available, then unmasked) BC thresholds obtained at the study visit and at the visit when the Ponto 4(s) was fitted. For subjects with SSD, AC thresholds on the non-implanted ear were used for this calculation.
Time Frame: Fitting Visit (at least 6 weeks prior to Study Visit 1 - data retrospectively collected) and Study Visit 1 (Day 1).
Population: MHL/CHL - n=11 SSD - n=5
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Ponto 4 Sound Processor Users
Number analyzed (Participants) | 16
dB
  MHL/CHL: number analyzed (Participants) | 11
  MHL/CHL | 0.114 (5.761)
  SSD: number analyzed (Participants) | 5
  SSD | 1.75 (2.88)

7. Secondary Outcome: J. To Assess if a Patient's With CHL/MHL Hearing Loss Has Degraded to Being Outside Fitting Range on the Implanted Ear(s).
Description: 1. BC hearing loss (PTA4), measured at the study visit, being outside intended fitting range (PTA4 >45 dB HL) compared to being inside fitting range (PTA<45 dB HL) at the time of the study visit.
Time Frame: fitting visit ≥6 weeks prior to study visit
Reporting Status: Not Posted, anticipated posting 2025-11

8. Secondary Outcome: K. To Asses if Patients' With CHL/MHL Air to Bone Gap (PTA4) Has Increased/Decreased on the Implanted Ear(s)
Description: 1. The difference between masked (if not available unmasked) BC and AC thresholds, denoted 'air to bone gap', calculated for frequencies 500, 1000, 2000 and 4000 Hz from audiogram measured at the study visit and the fitting visit.
Time Frame: Fitting Visit (at least 6 weeks prior to Study Visit 1 - data retrospectively collected) and Study Visit 1 (Day 1).
Population: Air to bone gap (PTA4) at fitting and study visit across MHL/CHL subjects.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Ponto 4 Sound Processor Users
Number analyzed (Participants) | 14
dB
  Fitting visit | 45.8 (13.6)
  Study visit | 50.2 (15.2)

9. Other Pre Specified Outcome: L. To Assess the Usage and Performance of Connectivity Device(s)
Description: 1. Questionnaire: Self-reported satisfaction ratings 0-10, for connectivity device(s) previously given to the test subject, where 0 is "very unsatisfied" and 10 is "very satisfied".
Time Frame: Visit 1, Day 1
Population: All participants included. Participants asked to rate their connectivity device(s) used, on a scale of 0.0 (very dissatisfied) to 10.0 (very satisfied).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ponto 4 Sound Processor Users
Number analyzed (Participants) | 19
units on a scale
  On App | 8.21 (2.10)
  Connect Clip | 6.90 (2.30)
  Remote Control | 8.00 (2.35)
  Edu Mic | 9.00 (0.00)

10. Other Pre Specified Outcome: F. To Assess the Usage Time With Ponto 4.
Description: Questionnaire: Self-reported usage hours per day during the month prior to the study visit across all subjects.
Time Frame: Visit 1, Day 1
Measure: Mean (Standard Deviation); unit: average hours/day
Arm/Group | Ponto 4 Sound Processor Users
Number analyzed (Participants) | 19
average hours/day | 12.6 (5.2)

11. Other Pre Specified Outcome: E. To Assess the Quality of Life of the Ponto 4
Description: GHSI Questionnaire: Scores across all subjects, on a scale from 0 to 100, with a higher score indicating a better quality of life.
Time Frame: Visit 1, Day 1 (For minors: Can be performed at a Visit 2, week 2, +/- 1 week)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Single Arm: Asessments for the hearing with Ponto 4 sound processor on the implanted ear(s).
  Audiometry: Audiometry: Thresholds from the audiogram obtained when Ponto 4 were fitted. Pure tone air conduction (AC) and bone conduction (BC) audiometry conducted at the visit.
  Speech recognition in quiet: Speech intelligibility is measured in a soundproof room using the Matrix sentences presented from a loudspeaker. The Matrix test includes five-word sentences with a fixed syntactical structure and limited contextual cues. A list of 20 sentences is compiled from these words, ensuring that no sentence is repeated twice. This test will be obtained both unaided and aided (with and without the Ponto 4(s)).
  Sound field Audiometry: Detection of sound field thresholds presented from a loudspeaker. Thresholds will be obtained both unaided and aided and the test order will be balanced between subjects. During these measurements, the Ponto 4 will be programmed in omni-directional mode, with noise reduction and feedback management system turned off.
Arm/Group | Single Arm
Number analyzed (Participants) | 19
units on a scale | 65.4 (11.7)

12. Other Pre Specified Outcome: D. To Assess the Subjective Experience of the Ponto 4
Description: SSQ Questionnaire: Scores across all subjects, on a subjective scale from 0-10, where 0 is "the worst" and 10 is "the best"
Time Frame: Visit 1,Day 1 (For minors: Can be performed at a Visit 2, week 2, +/- 1 week)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 19
units on a scale | 6.28 (1.91)

ADVERSE EVENTS:
Time Frame: study duration was one, approximately 2 hour long, visit.
Description: No adverse events nor device deficiencies were encountered during the study. No serious adverse events were encountered during the study.
Groups:
- Ponto 4 Sound Processor Users: Assessments of users with Ponto 4 sound processor on the implanted ear(s).
Arm/Group | Ponto 4 Sound Processor Users
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT04761926/Prot_SAP_000.pdf